CLINICAL TRIAL: NCT01759472
Title: Effect of Montelukast on Leukotriene Sensitive Asthma Detected by LTD4 Bronchial Provocation Test
Brief Title: Effect Study of Montelukast to Treat Asthma Detected by LTD4 Bronchial Effect Study of Montelukast to Treat Asthma Detected by LTD4 Bronchial Provocation Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Xu Shi, Guangzhou Institute of Respiratory Disease, Guangzhou Institute of Respiratory Disease
Other Study IDs: 2012BAI05B01
Record Dates: First submitted 2012-12-28; First posted 2013-01-03 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Bronchial Asthma
Keywords: leukotriene; leukotriene receptor antagonist
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- montelukast，vitamin C pill: leukotriene receptor antagonist:(montelukast)，montelukast (10 mg, once per night)，56 days vitamin C pill:100mg，once per night，56 days
- montelukast, vitamin C pill: montelukast:10 mg, once per night，56 days vitamin C pill:100mg，once per night，56 days

SUMMARY:
To determine whether LTD4-BPT could be an effective indicator for predicting efficacy of anti-leukotriene therapy, allowing objective proofs for the use of LTRA among asthmatics in a specific sensitive to leukotriene population of asthma.

Hypothesis ：Monteluakst can better improve pre-challenge FEV1 from baseline in leukotriene-sensitive group than leukotriene-insensitive group.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 15-60 years, male or female.
2. Mild to moderate persistent asthma.
3. Mini AQLQ score ≤6 or ACQ score ≥1.
4. Giving written informed consent.

Exclusion Criteria:

1. Current smoker or quitted smoking ≤12 months.
2. Significant allergen exposure.
3. Respiratory tract infection within 2 weeks before or during the study.
4. Cardiovascular disease.
5. History of malignant disease within the preceding 5 years.
6. And/or concomitant pulmonary disease.
7. Pregnant or breast-feed period.
8. Use of leukotrienes receptor antagonist within 5 days

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Bronchial Asthma patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
whether there was improvement in pre-challenge FEV1% | from commencement of LTRA therapy to (7±2) days and (56±5) days
  The primary outcome was a qualitative measure, with the results being expressed as either yes or no ('1' or '0' in Logistic model).A higher FEV1% is more suggestive of instability of asthma control.

SECONDARY OUTCOMES:
whether there was improvement in post- treatment FENO | from commencement of LTRA therapy to (7±2) days and (56±5) days
  In Logistic regression model, whether there was improvement shown in post-treatment FENO as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure was qualitative one. FENO represented fractional exhaled nitric oxide above.

OTHER OUTCOMES:
whether there was improvement in post- treatment PD20FEV1-MCH | from commencement of LTRA therapy to (7±2) days and (56±5) days
  In Logistic regression model, whether there was improvement shown in post-treatment PD20FEV1-MCH as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure above was qualitative. PD20FEV1-MCh referred to as the provocative dosage causing a 20% fall in FEV1 while using methacholine as a bronchoprovocant.
whether there was improvement in post- treatment AQLQ symptom score | from commencement of LTRA therapy to (7±2) days and (56±5) days
  In Logistic regression model, whether there was improvement shown in post-treatment AQLQ symptom score as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure above was qualitative. Items with regard to asthma symptoms were extracted from the whole AQLQ score, with the total score of 84. Higher score represented better asthma control.
whether there was improvement in post- treatment ACT score | from commencement of LTRA therapy to (56±5) days
  In Logistic regression model, whether there was improvement shown in post-treatment ACT score as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure above was qualitative. The total score of ACT was 25, with 5 questions in all. Higher score was indicative of better asthma control.
whether there was a gradual decrease in weekly use of salbutamol | from commencement of LTRA therapy to (56±5) days
  In Logistic regression model, whether there was a gradual decrease in weekly use of salbutamol as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure was qualitative one.
improvement in weekly and monthly PEFR | from commencement of LTRA therapy to (56±5) days
  The primary outcome was a qualitative measure, with the results being expressed as either yes or no ('1' or '0' in Logistic model).PEFR was defined as the changed rate of peak expiratory flow, which was calculated using the formula according to maximal PEF (PEFmax) and minimal PEF (PEFmin) measured by portable PEF monitor: 100%*(PEFmax-PEFmin)/[(PEFmax+PEFmin)*1/2]. A higher PEFR is more suggestive of instability of asthma control.
whether there was improvement in post- treatment PD20FEV1-LTD4 | from commencement of LTRA therapy to (7±2) days and (56±5) days
  In Logistic regression model, whether there was improvement shown in post-treatment PD20FEV1-LTD4 as compared with pre-treatment level was expressed as either 'yes' or 'no', with symbols of '1' or '0'. Thus the measure above was qualitative. PD20FEV1-LTD4 referred to as the provocative dosage causing a 20% fall in FEV1 while using Leukotriene D4 as a bronchoprovocant.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, State Key Laboratory of Respiratory Disease, Guangzhou, Guangdong, China